CLINICAL TRIAL: NCT02035228
Title: Abdominal Functional Electrical Stimulation to Reduce Hyperinflation in Patients With Chronic Obstructive Pulmonary Disease: A Feasibility Study
Brief Title: Abdominal Functional Electrical Stimulation to Reduce Hyperinflation in Chronic Obstructive Pulmonary Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liberate Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: LM-SB-001
Record Dates: First submitted 2014-01-10; First posted 2014-01-14 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic Obstructive Pulmonary Disease; Lung Hyperinflation; Abdominal Muscle; Functional Electrical Stimulation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Seated (Experimental): Patients breathing will be compared across a series of 9 trials in which unassisted breathing is compared to abdominal stimulation (SecondBreath) assisted breathing at various intensities. Each breathing trial will last for 2 minutes and will be conducted while the patient is seated. The following abdominal stimulation trials were included:
  Abdominal Stimulation - low / early Abdominal stimulation - low/late Abdominal Stimulation - low/full Abdominal stimulation - med/early Abdominal stimulation - med/late Abdominal Stimulation - med/full Abdominal Stimulation - high/early Abdominal Stimulation - high/late Abdominal Stimulation - high/full
  Interventions: Device: Abdominal Stimulation - low / early; Device: Abdominal stimulation - low/late; Device: Abdominal Stimulation - low/full; Device: Abdominal stimulation - med/early; Device: Abdominal stimulation - med/late; Device: Abdominal Stimulation - med/full; Device: Abdominal Stimulation - high/early; Device: Abdominal Stimulation - high/late; Device: Abdominal Stimulation - high/full
- 6 minute step test (Experimental): Patients will complete a 6 minute step test with and without abdominal stimulation (SecondBreath).
  Abdominal Stimulation - high/full
  Interventions: Device: Abdominal Stimulation - high/full

INTERVENTIONS:
Device: Abdominal Stimulation - low / early — Transcutaneous electrical stimulation applied to the abdominal wall muscles in synchronous with volitional exhalation.
  Stimulation is applied at low stimulation current for the first half of exhalation
  Other Names: SecondBreath
  Arms: Seated
Device: Abdominal stimulation - low/late — Transcutaneous electrical stimulation applied to the abdominal wall muscles in synchronous with volitional exhalation.
  Stimulation is applied at low stimulation current for the second half of exhalation
  Other Names: SecondBreath
  Arms: Seated
Device: Abdominal Stimulation - low/full — Transcutaneous electrical stimulation applied to the abdominal wall muscles in synchronous with volitional exhalation.
  Stimulation is applied at low stimulation current throughout exhalation
  Other Names: SecondBreath
  Arms: Seated
Device: Abdominal stimulation - med/early — Transcutaneous electrical stimulation applied to the abdominal wall muscles in synchronous with volitional exhalation.
  Stimulation is applied at medium stimulation current for the first half of exhalation
  Other Names: SecondBreath
  Arms: Seated
Device: Abdominal stimulation - med/late — Transcutaneous electrical stimulation applied to the abdominal wall muscles in synchronous with volitional exhalation.
  Stimulation is applied at medium stimulation current for the second half of exhalation
  Other Names: SecondBreath
  Arms: Seated
Device: Abdominal Stimulation - med/full — Transcutaneous electrical stimulation applied to the abdominal wall muscles in synchronous with volitional exhalation.
  Stimulation is applied at medium stimulation current throughout exhalation
  Other Names: SecondBreath
  Arms: Seated
Device: Abdominal Stimulation - high/early — Transcutaneous electrical stimulation applied to the abdominal wall muscles in synchronous with volitional exhalation.
  Stimulation is applied at high stimulation current for the first half of exhalation
  Other Names: SecondBreath
  Arms: Seated
Device: Abdominal Stimulation - high/late — Transcutaneous electrical stimulation applied to the abdominal wall muscles in synchronous with volitional exhalation.
  Stimulation is applied at hig stimulation current for the second half of exhalation
  Other Names: SecondBreath
  Arms: Seated
Device: Abdominal Stimulation - high/full — Transcutaneous electrical stimulation applied to the abdominal wall muscles in synchronous with volitional exhalation.
  Stimulation is applied at high stimulation current throughout exhalation
  Other Names: SecondBreath

SUMMARY:
This is an early feasibility study to investigate whether transcutaneous electrical stimulation applied to the abdominal wall muscles synchronous with voluntary exhalation can be used to support ventilation and affect hyperinflation in patients with chronic obstructive pulmonary disease. As part of this study, the effect of a range of stimulation intensities and stimulation timing profiles will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Post-bronchodilator FEV1/FVC ratio of less than 0.7 and post-bronchodilator FEV1 between 30 and 80 % predicted.
* Current or former smokers with at least a 20 pack year smoking history
* Over the age of forty

Exclusion Criteria:

* Female subjects who are pregnant
* Subjects unable to give informed consent
* Subjects unable to perform required activities of the study (e.g. Six minute walk test)
* Subjects with an implanted electronic device (e.g. a cardiac pacemaker)
* Subjects who have had a chronic obstructive pulmonary disease exacerbation within 30 days prior to enrollment
* Considerable arthritic changes that limit exertion
* Patients on oral prednisone
* Patients with a hernia
* Patients with a history of pneumothorax within the last 5 years
* History of epilepsy
* History of Abnormal electrocardiogram suggestive of cardiac disease

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change in inspiratory capacity during 2 minutes of resting breathing when patients were seated | 2 minutes
  Inspiratory Capacity was measured before and after two minute periods of volitional and abdominal stimulation assisted breathing. The two minute trials of breathing were measured while patients were seated.
Change in inspiratory capacity during a 6 minute step test | 6 minutes

SECONDARY OUTCOMES:
Average tidal volume during 2 minutes of resting breathing while seated | 2 minutes
Average minute ventilation during 2 minutes of resting breathing while seated | 2 minutes
Average peak expiratory flow rate during 2 minutes of resting breathing while seated | 2 minutes
Average breathing rate during two minutes of resting breathing while seated | 2 minutes
Change in dyspnea measured using the modified Borg dyspnea scale during a 6 minute step test | 6 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Rodney Folz, PhD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States